CLINICAL TRIAL: NCT03281915
Title: Comparison Between Impact of Inguinal and Subinguinal Approaches of Varicocelectomy on Semen Parameters in Patients With Normal Semen Analysis
Brief Title: the Effect of Different Modialites of Varicocelectomy on Semen Parameters in Patient With Normal Semen Analysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Abdelkader, Resident, Assiut University
Other Study IDs: varicocelectomy
Record Dates: First submitted 2017-08-25; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Varicocele
Keywords: infertility; pain; pregnancy
MeSH Terms: conditions — Varicocele; Infertility; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high inguinal approch: Patients undergoing high inguinal varicocelectomy with normal pre operative semen parameters, post operative semen analysis parameters will be recorded
  Interventions: Procedure: High inguinal Varicocelectomy
- subinguinal approch: Patients undergoing subinguinal varicocelectomy with normal pre operative semen parameters, post operative semen analysis parameters will be recorded
  Interventions: Procedure: Subinguinal varicocelectomy

INTERVENTIONS:
Procedure: High inguinal Varicocelectomy — Semen parameters after high inguinal varicocelectomy will be collected
  Groups: high inguinal approch
Procedure: Subinguinal varicocelectomy — Semen parameters after subinguinal Varicocelectomy will be collected
  Groups: subinguinal approch

SUMMARY:
to evalute the effect inguinal and subinguinal approach of varicoceclectomy on semen parameter for patients complaining of varicocele with normal semen parameter (pain is the main complaint)

DETAILED DESCRIPTION:
the varicocele is defined as dilated and incompetent veins within the pampiniform plexus of spermatic cord. varicocele has been described as the most common surgically correctable cause of male subinfertility.this is a disease that devolops during puberty when both endocrine and exocrine function of the testicle dramatically increases, along with testicular blood flow. varicocele only rarely detected in boys less than 10 years. left sided varicocle found in 15% of healthy young men.incontrast, the incidence in sub fertile men approaches 40% bilateral varicocele is uncommon in healthy men (less than 10%) but palpated in 20% in sub fertile men. in-general varicocele don't spontaneously regress. an accurate physical examination remain the corner stone of varicocele diagnosis.

several anatomic features contribute to the predominance of left sided varicocele is the left intrnal spermatic vein longer than the right and it typically joins the left renal vein at a right angle.as result of this character higher venous pressures fair transmited to the left spermatic vein and result in reterograde reflux of blood.

varicocle are associated with testicular atrophhy and varicocle correction can reverse atrophy in adolececnt. there is strong evidence affect semen quality it can cause abnormalties in concentration, motility and morphology.main defect is the motility.

indication of varicocelectomy:

1. Large varicoceles in adolescents
2. Childhood varicocele with testicular atrophy
3. Varicoceles with elevated FSH values, or low testosterone levels
4. Varicoceles with scrotal pain
5. Cosmetic indication
6. Male infertility with pathological semen analysis and varicocele

ELIGIBILITY:
Inclusion Criteria:

* age more than 19 years old
* primary varicocele

Exclusion Criteria:

* secondary varicocele recurrent varicocele age less than 19 years

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Male patients undergoing varicocelectomy while having normal semen parameters (doing surgery for other reasons eg. pain)
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2017-10-15 (Estimated); Primary Completion 2018-10-15 (Estimated); Study Completion 2018-10-15 (Estimated)

PRIMARY OUTCOMES:
Semen analysis | 3months
  Motility morphology concentration

CONTACTS AND LOCATIONS:
Overall Officials: Ehab O Ahmed, Study Director — unaffiliation; Mohamed I Taha, Study Chair — unaffiliation; Ahmed k mohamed, Study Director — unaffiliation
Locations (1):
- Assuit Medical School, Asyut, Assuit, Egypt

REFERENCES:
- [Background] Leslie SW, Sajjad H, Siref LE. Varicocele. 2023 Nov 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448113/ PMID 28846314
- [Background] Wu X, Liu Q, Zhang R, Wang W, Gao Y. Therapeutic efficacy and safety of laparoscopic surgery versus microsurgery for varicocele of adult males: A meta-analysis. Medicine (Baltimore). 2017 Aug;96(34):e7818. doi: 10.1097/MD.0000000000007818. PMID 28834886
- [Background] Canning DA. Re: Sperm Concentration and Forward Motility are Not Correlated with Age in Adolescents with an Idiopathic Varicocele and Symmetrical Testicular Volumes. J Urol. 2017 Sep;198(3):472. doi: 10.1016/j.juro.2017.06.068. Epub 2017 Jun 20. No abstract available. PMID 28817895
- [Background] Schmidt B. Membranes in artificial organs. Artif Organs. 1996 May;20(5):375-80. doi: 10.1111/j.1525-1594.1996.tb04519.x. PMID 8725614
- [Background] Sedaghatpour D, Berookhim BM. The Role of Varicocele in Male Factor Subfertility. Curr Urol Rep. 2017 Sep;18(9):73. doi: 10.1007/s11934-017-0713-8. PMID 28718159